CLINICAL TRIAL: NCT05553769
Title: Physiological Adaptations to Resistance Training, Detraining, and Retraining in Young Healthy Males and Females
Brief Title: Resistance Training, Detraining, and Retraining Study 2022
Acronym: TraDeRe2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TraDeRe2022
Record Dates: First submitted 2022-03-02; First posted 2022-09-23 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Exercise Training; Skeletal Muscle; Skeletal Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants (healthy untrained men and women, age 18-40) start with a 3-week familiarization and baseline measurement period. After that, they are randomized to two intervention groups, where other group will conduct 10-week RT intervention and a 10-week DT period and again the exact same 10-week RT intervention again whereas the other group start with a 10-week non-training period and then continues with a 20-week RT intervention. RT consists of two training sessions per week of total body workouts. Same measurements are conducted for both groups with the same time intervals.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 week training, 10 week detraining, 10 week retraining (Experimental): Participants (healthy untrained men and women, age 18-40) will conduct 10-week RT intervention and a 10-week DT period and the exact same 10-week RT intervention again. RT consists of two training sessions per week of total body workouts.
  Interventions: Other: Resistance training, detraining, retraining
- 10 week non-training, 20 week continuous training (Experimental): Participants (healthy untrained men and women, age 18-40) start with a 10-week non-training period and then continues with a 20-week RT intervention. RT consists of two training sessions per week of total body workouts.
  Interventions: Other: Resistance training, detraining, retraining

INTERVENTIONS:
Other: Resistance training, detraining, retraining — Participants (healthy untrained men and women, age 18-40) start with a 3-week familiarization and baseline measurement period. After that, they are randomized to two intervention groups, where other group will conduct 10-week RT intervention and a 10-week DT period and again the exact same 10-week RT intervention again whereas the other group start with a 10-week non-training period and then continues with a 20-week RT intervention. RT consists of two training sessions per week of total body workouts. Same measurements are conducted for both groups with the same time intervals.

SUMMARY:
The research project is aiming to examine the muscular adaptations to resistance training (RT), detraining (DT) and repeated RT (i.e. retraining). The research project will also examine differences in muscular adaptations between 20 weeks of continuous RT and 20 weeks of intermittent RT including a 10-week DT period in the middle of the training intervention. This is randomized controlled trial in which the research participants will be randomized into discontinuous and continuous groups (both n=~20). Both will be doing a 2-3-week familiarization and control period at the start. Then in the former there will be an initial strength training period (10-wks), a DT period (10-wks), and a second strength training (retraining) period (10-wks). The second group includes a 10-wk non-training control period (10-wks) followed by a RT period (20-wks). Participants will be young, healthy men and women (age 18-35, which 50% are females) with no systematic RT experience during the last 6 months. Measurements will be completed before and after each study period. Body composition will be measured via bioelectrical impedance analysis (BIA) and 3D body scans. Dynamic leg press and elbow flexion one repetition-maximum (1RM) will be used to test maximal strength. Anaerobic performance and strength endurance will be tested in elbow flexion and dynamic leg press using RM tests. Vastus lateralis (VL) and biceps brachii muscle cross-sectional area (CSA) will be assessed via ultrasound. Muscle biopsies of the VL muscle will be obtained to assess changes in muscle fiber morphology and factors regulating and associated with the hypertrophic processes and metabolism. Blood samples will be collected to analyze changes in metabolism and physiology. A rating of perceived exertion (RPE) during training will be collected after every exercise to ensure proper training intensity. Finally, nutrition and habitual physical activity will be assessed with 4-day diet diaries and physical activity questionnaires before the intervention and during each 10-week period.

DETAILED DESCRIPTION:
It is well known that RT increases skeletal muscle size and strength. However, there seems to be a difference in increases in muscle size (termed hypertrophy) and strength in upper and lower limb musculature in untrained population after RT. Moreover, there is large inter-individual variation in the adaptations gained through RT. Also at the moment, the responses to de- and retraining are not well known, and new research designs for investigating possible muscle memory are needed. Muscle mass and strength, once achieved with RT, can be obtained faster with subsequent retraining if the initial adaptations were lost due to inactivity. RT causes many molecular and cellular changes in myofibers that aid in hypertrophic processes, yet their adaptations to DT and contribution to muscle memory are still marginally researched. It is, therefore, essential to widen our knowledge about the permanence of physiological adaptations in skeletal muscle to periods of DT and repeated exposure to RT.

The primary objectives to achieve by this project are:

1. to determine the magnitude of 10-week RT period on upper and lower limb maximal dynamic strength and muscle size compared to the non-training control group
2. to determine whether the responses to 20-week continuous RT differs in adaptations in maximal strength and muscle hypertrophy from two 10-week RT periods separated by a 10-week detraining period
3. to identify molecular and cellular biomarkers explaining responses to RT, detraining and retraining

ELIGIBILITY:
Inclusion Criteria:

* No regular resistance training history
* BMI within range 18.5-30 kg/m2
* Participants must be 18-40 years old
* No history in systematic endurance-type training (> 2 endurance exercise sessions lasting > 30 minutes per week for the last six months)
* non-smoker
* not currently consuming any anti-inflammatory drug(s)

Exclusion Criteria:

* history of medication that could affect exercise responses
* use of nutritional supplements aside from those that are protein- or carbohydrate-based (ex. creatine) or basic minerals, vitamins, or fish oil products
* any acute or chronic illness affecting cardiovascular, respiratory, musculoskeletal and/or endocrine function
* any other condition that may limit the ability to perform resistance training and testing (ex. uncontrolled hypertension, diabetes, arthritic conditions, neuromuscular complications)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in upper and lower limb maximal strength after 10-week RT | week -2, week 0, week 10
  Maximal muscle strength will be assessed via one repetition maximum (1RM) tests of both the leg press and barbell biceps curl exercises according to the NSCA's guidelines.

SECONDARY OUTCOMES:
Change in muscular performance after 20-week continuous RT period and two 10-week RT periods separated by a 10-week DT period | week -2, week 0, week 10, week 20, week 30
  Change in 1 repetition maximum and 10 repetition maximum tests in dynamic leg press and biceps curl exercises, maximal force in isometric knee extension test, and flight time in countermovement jump.
Change in upper and lower limb muscle CSA after 10-week RT period | week -2, week 0, week 10
  Vastus lateralis and biceps brachii muscle cross-sectional area (mm2) and thickness (mm) at the mid-limb will be assessed using a B-mode axial plane ultrasound (model SSD-α10, Aloka, Tokyo, Japan) with a 10 MHz linear-array probe (60 mm width) in extended-ﬁeld-of-view mode (23 Hz sampling frequency).
Change in upper and lower limb muscle CSA after 20-week continuous RT period and two 10-week RT periods separated by a 10-week DT period | week 0, week 10, week 20, week 30
  Vastus lateralis and biceps brachii muscle cross-sectional area (mm2) and thickness (mm) at the mid-limb will be assessed using a B-mode axial plane ultrasound (see above).
Changes in muscle fiber size during the intervention period | week 0, week 10, week 20, week 30
  Vastus lateralis muscle biopsy
Change in lean mass during the intervention period | week -2, week 0, week 10, week 20, week 30
  BIA (InBody 770, Biospace Co. Seoul, Korea) method will be utilized to estimate changes in lean mass (kg).
Change in fat mass during the intervention period | week 0, week 10, week 20, week 30
  BIA (InBody 770, Biospace Co. Seoul, Korea) method will be utilized to estimate changes in fat mass (kg).
Change in body segment volumes during the intervention period | week 0, week 10, week 20, week 30
  3Dscanning (Fit3D, USA) will be used to estimate upper and lower limb body segment volumes (cm3).

OTHER OUTCOMES:
Changes in muscle fiber morphology and metabolism during the intervention period | week 0, week 10, week 20, week 30
  Change in muscle fiber cross-sectional area, fiber type, mitochondrial count, and capillary density will be determined by immunohistochemistry. Anaerobic enzymes and sarcoplasmic protein contents in myofibers will be measured by Western blotting and by SDS-PAGE.
Changes in metabolomics during the intervention period | week 0, week 10, week 20, week 30
  A high-throughput serum Nuclear Magnetic Resonance (NMR) metabolomics platform will be used for the absolute quantification of serum lipids and metabolite profile. The NMR metabolome assay yields at least 220 different metabolites including amino acids, apolipoproteins, cholesterol, fatty acids, glycolysis related metabolites, and inflammation markers. Serum metabolomics will be quantified from acquired fasting blood samples by Nightingale (Finland) company, specializing in metabolomics quantification. Further, statistical analysis of provided data will be handled at Finnish Institute for Health and Welfare (THL, Finland). In addition, mass spectrometry based targeted/untargeted metabolomics analysis will be conducted from serum and/or muscle samples if funding for those analysis is available.
Changes in proteomics during the intervention period | week 0, week 10, week 20, week 30
  From muscle samples, we harness the advanced capabilities of DIA-PASEF (Data-Independent Acquisition Parallel Accumulation Serial Fragmentation) on the cutting-edge timsTOF Pro LC-MS platform to enable deep proteomics analysis. The analysis happens in our collaborators Dr. Varjosalo´s laboratory in the University of Helsinki, Finland. By integrating DIA-PASEF's unparalleled efficiency in ion fragmentation and parallel accumulation with the high-resolution mass spectrometry of timsTOF Pro, we anticipate a remarkable increase in the number and quality of protein identifications from muscle cells.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jyväkylä, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halonen EJ, Gabriel I, Kelahaara MM, Ahtiainen JP, Hulmi JJ. Does Taking a Break Matter-Adaptations in Muscle Strength and Size Between Continuous and Periodic Resistance Training. Scand J Med Sci Sports. 2024 Oct;34(10):e14739. doi: 10.1111/sms.14739. PMID 39364857